CLINICAL TRIAL: NCT06922994
Title: Statin Effect on Arrhythmogenic Cardiomyopathy Disease Progression
Brief Title: Statin Effect on Arrhythmogenic Cardiomyopathy Disease Progression (SEARCH)
Acronym: SEARCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Federico II University (Other); Università Politecnica delle Marche (Other); Ospedali dei Colli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEARCH; PNRR-MCNT2-2023-12376978 (Other Grant/Funding Number: European Union - NextGenerationEU); 2024-514643-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-20; First posted 2025-04-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-04

CONDITIONS: Arrhythmogenic Cardiomyopathy
Keywords: Atorvastatin; Strain; Disease progression risk; Arrhythmias
MeSH Terms: conditions — Sprains and Strains; Arrhythmias, Cardiac | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized, clinical study: Atorvastatin 80mg/day or placebo will be administered for 18 months to 102 ACM patients, and the endpoints will be tested.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Active Comparator): Atorvastatin arm will be composed by 51 patients affected by Arrhythmogenic Cardiomyopathy.
  Interventions: Drug: Atorvastatin 80 mg/day
- Placebo (Placebo Comparator): Placebo arm will be composed by 51 patients affected by Arrhythmogenic Cardiomyopathy.
  Interventions: Drug: Placebo atorvastatin

INTERVENTIONS:
Drug: Atorvastatin 80 mg/day — Atorvastatin 80mg/day will be administered for 18 months to patients affected by Arrhythmogenic Cardiomyopathy
  Arms: Atorvastatin
Drug: Placebo atorvastatin — One tablet of placebo will be administered for 18 months to patients affected by Arrhythmogenic Cardiomyopathy
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Atorvastatin 80 mg is effective to avoid functional right ventricular deterioration in patients affected by Arrhythmogenic Cardiomyopathy. It will also learn about the safety of Atorvastatin 80 mg in this type of patients. The main questions it aims to answer are:

1. Does Atorvastatin 80 mg prevent worstening of the right ventricular functioning?
2. Does Atorvastatin 80 mg prevent the worsening of electric, morphological and biomarkers deterioration?
3. What medical problems do participants have when taking Atorvastatin 80 mg?

Researchers will compare Atorvastatin 80 mg to a placebo (a look-alike substance that contains no drug) to see if the drug works to treat Arrhythmogenic Cardiomyopathy.

Participants will:

1. Take Atorvastatin 80 mg or a placebo every day for 18 months;
2. Visit the clinic at the enrollment and after 2, 4, 9 and 18 months for checkups and tests;
3. Make a phone call for safety check after 12, 15 and 19 months since the enrollment;
4. Fill out psychological questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age, at the time of signing the informed consent
2. Participants affected by Arrhythmogenic Cardiomyopathy as defined by task force criteria

Exclusion Criteria:

1. Known hypersensitivity to atorvastatin or any of the excipients
2. Moderate or severe liver disease
3. Muscle disease
4. Left ventricular ejection fraction <35%
5. Congestive heart failure defined by the New York Heart Association (NYHA) as class III or IV.
6. Known cardiomyopathy of other origin: post ischemic, hypertrophic, idiopathic dilated, restrictive; known moderate-to-severe mitral or aortic valvulopathy; pulmonary hypertension; congenital cardiac abnormalities
7. Hypercholesterolemic patients that require the use of lipid lowering drugs.
8. Heart transplantation
9. Estimated life expectancy of less than 2 years
10. Any other medical condition that, in the judgment of the investigator, places the patient at risk or makes the patient unreliable or limits the patient's ability to complete the study
11. Potent CYP3A4 modifiers such as Erythromycin, Clarithromycin Azole antifungals, Protease inhibitors , Gemfibrozil, Ciclosporin, Danazol
12. Fusidic acid (drug for bacterial infections)
13. Hepatitis C antivirals as telaprevir, boceprevir, glecaprevir/pibrentasvir and ledipasvir/sofosbuvir combination
14. Any other lipid lowering drugs such as Statins, Cholesterol absorption inhibitors, Bile acid sequestrants , PCSK9 inhibitors, Adenosine triphosphate-citrate lyase inhibitors , Fibrates, Omega-3 fatty acid ethyl esters
15. Drugs primary indicated as antioxidants
16. Enrollment in another clinical trial or past clinical trial in which an investigational drug was administered within 30 days of Visit 1 or within the 5 half-lives of the investigational drug, whichever is longer.
17. Pregnant or lactating women
18. Women of childbearing age who are not using adequate contraception
19. Known dependency on alcohol - drug abuse.
20. Contraindications to cardiac magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Atorvastatin in avoiding functional right ventricular deterioration | From enrollment to the end of treatment at 18 months
  Variation of right ventricular free wall longitudinal strain measured by echocardiography after 18 months respect to baseline (%)

SECONDARY OUTCOMES:
Safety of Atorvastatin treatment | From enrollment to 1 month after the end of treatment (19 months)
  Monitoring of adverse events and patient's well-being.
Efficacy of Atorvastatin in avoiding morphological deterioration (ventricular volumes) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of other morphological parameters measured both at echocardiography and cardiac magnetic resonance: ventricular volumes (ml)
Efficacy of Atorvastatin in avoiding morphological deterioration (wall thickness ) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of other morphological parameters measured both at echocardiography and cardiac magnetic resonance: wall thickness (mm)
Efficacy of Atorvastatin in avoiding morphological deterioration (cardiac function ) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of other morphological parameters measured both at echocardiography and cardiac magnetic resonance: cardiac function (%)
Efficacy of Atorvastatin in avoiding arrhythmic deterioration (premature ventricular contractions) | From enrollment to the end of treatment at 18 months
  Deterioration from baseline of arrhythmia burden: premature ventricular contractions (number in the 24h)
Efficacy of Atorvastatin in avoiding arrhythmic deterioration (nonsustained ventricular arrhythmias) | From enrollment to the end of treatment at 18 months
  Deterioration from baseline of arrhythmia burden: nonsustained ventricular arrhythmias (number)
Efficacy of Atorvastatin in avoiding arrhythmic deterioration (sustained ventricular arrhythmias) | From enrollment to the end of treatment at 18 months
  Deterioration from baseline of arrhythmia burden: sustained ventricular arrhythmias (number)
Efficacy of Atorvastatin in avoiding arrhythmic deterioration (ventricular fibrillation ) | From enrollment to the end of treatment at 18 months
  Deterioration from baseline of arrhythmia burden: ventricular fibrillation (number)
Efficacy of Atorvastatin in avoiding arrhythmic deterioration (ICD shocks) | From enrollment to the end of treatment at 18 months
  Deterioration from baseline of arrhythmia burden: appropriate ICD shocks (number)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (QRS) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: QRS duration (ms)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (QT) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: QT duration (ms)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (PR) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: PR duration (ms)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (amplitudes) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: amplitude of the potential (mV)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (T wave) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: ), T wave inversion (number of presences in V1-V6)
Efficacy of Atorvastatin in avoiding electrocardiographic deterioration (ԑ wave) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of electrocardiographic parameters: ԑ wave in V1-V3 (presence)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (oxLDL) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: oxLDL (mU/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (MDA) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: MDA (ng/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (4HNE) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: 4HNE (pg/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (estradiol) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: estradiol (pg/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (testosterone) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: testosterone (ng/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (BIN1) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: BIN1 (pg/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (GAL3) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: GAL3 (ng/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (HSP70) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: HSP70 (ng/mL)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (TGFb) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: TGFb (pg/mL)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (ST2) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: ST2 (ng/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (BNP) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: BNP (pg/mL)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (NTproBNP) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: NTproBNP (pg/mL)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (hs-cTnI) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: hs-cTnI (ng/L)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (CRP) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: CRP (mg/L)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (IL6) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: IL6 (pg/ml)
Efficacy of Atorvastatin in avoiding biomarkers deterioration (TNF alfa) | From enrollment to the end of treatment (18 months)
  Deterioration from baseline of blood parameters: TNF alfa (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Tondo, Principal Investigator — Centro Cardiologico Monzino IRCCS
Locations (5):
- Italy (5):
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia, PV
  - Università Politecnica delle Marche, Ancona
  - Centro Cardiologico Monzino IRCSS, Milan
  - AORN - Ospedali dei Colli, Napoli
  - Università degli Studi di Napoli Federico II, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommariva E, Stadiotti I, Casella M, Catto V, Dello Russo A, Carbucicchio C, Arnaboldi L, De Metrio S, Milano G, Scopece A, Casaburo M, Andreini D, Mushtaq S, Conte E, Chiesa M, Birchmeier W, Cogliati E, Paolin A, Konig E, Meraviglia V, De Musso M, Volani C, Cattelan G, Rauhe W, Turnu L, Porro B, Pedrazzini M, Camera M, Corsini A, Tondo C, Rossini A, Pompilio G. Oxidized LDL-dependent pathway as new pathogenic trigger in arrhythmogenic cardiomyopathy. EMBO Mol Med. 2021 Sep 7;13(9):e14365. doi: 10.15252/emmm.202114365. Epub 2021 Aug 2. PMID 34337880